CLINICAL TRIAL: NCT06306339
Title: A Phase 2a Multi-center, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Efficacy and Safety of Burfiralimab(hzVSF-v13) Added to Disease-modifying Antirheumatic Drugs in Participants With Moderate to Severe RA
Brief Title: A Study to Assess the Efficacy and Safety of Burfiralimab (hzVSF-v13) and DMRD (Disease-modifying Antirheumatic Drug)
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: ImmuneMed, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: hzVSF_v13-0015
Record Dates: First submitted 2024-02-07; First posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-02

CONDITIONS: Moderate to Severe Rheumatoid Arthritis
Keywords: Rheumatoid arthritis, RA
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo infusion (Placebo Comparator): Placebo + SOC
  Interventions: Drug: SOC (Standard of care); Drug: Placebo
- Burfiralimab(hzVSF-v13) 200mg IV infusion (Experimental): Burfiralimab (hzVSF-v13) 200mg/dose + SOC
  Interventions: Drug: Burfiralimab; Drug: SOC (Standard of care)
- Burfiralimab(hzVSF-v13) 600mg IV infusion (Experimental): Burfiralimab (hzVSF-v13) 600mg/dose + SOC
  Interventions: Drug: Burfiralimab; Drug: SOC (Standard of care)

INTERVENTIONS:
Drug: Burfiralimab — Humanized monoclonal antibody.
  Other Names: hzVSF-v13
  Arms: Burfiralimab(hzVSF-v13) 200mg IV infusion; Burfiralimab(hzVSF-v13) 600mg IV infusion
Drug: SOC (Standard of care) — The following medications listed are allowed to be administered during the course of the clinical study.
  1. biologic disease-modifying antirheumatic drug (bDMARD)
  2. conventional synthetic disease-modifying antirheumatic drug (csDMARD)
  Other Names: bDMARD or csDMARD
Drug: Placebo — The placebo for Burfiralimab (hzVSF-v13)
  Other Names: The placebo for Burfiralimab (hzVSF-v13)
  Arms: Placebo infusion

SUMMARY:
The goal of this clinical trial is to evaluate the efficacy and safety of intravenous infusions of burfiralimab (hzVSF-v13) when added to Disease-Modifying Antirheumatic Drug (DMARD) treatment as Standard of Care (SOC) in participants with moderate to severe Rheumatoid Arthritis (RA).

DETAILED DESCRIPTION:
This study is a Phase 2a, multi-center, randomized, double-blind, placebo-controlled. Efficacy and safety of biweekly intravenous infusions of burfiralimab (hzVSF-v13), added to DMARD treatment as standard of care, is evaluated in comparison with placebo. Participants of either sex, aged, 18~80years, are enrolled it they have moderate to severe RA and had an inadequate response to disease-modifying antirheumatic drug(DMARD) treatments. The study consists of a screening period for up to 4 weeks, a treatment period of 10 weeks. Eligible participants are randomized in a 1:1:1 ratio to 1 of the 3 treatment groups: 200mg burfiralimab (hzVSF-v13) + SOC (study group 1), 600mg burfiralimab (hzVSF-v13) + SOC (study group 2), or placebo + SOC (control group). The primary focus of the study is to evaluate preliminary of the 2 doses of burfiralimab (hzVSF-v13, 200mg to 600mg) administered by IV infusion biweekly for 10 weeks when compared to placebo in lowering disease activity in participants. Efficacy analyses evaluate disease and health-related quality of life improvements at week 12 and week 18. Safety is assessed at up to 18 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Participant has a diagnosis of adult-onset RA for at least 3 months prior to Screening, as defined by the 2010 ACR/European League Against Rheumatism (EULAR) classification criteria.
2. Participant has moderate to severe RA at Screening and Baseline.
3. Participant has had an inadequate response to, loss of response, or intolerance to at least 2 bDMARDs or tsDMARDs.
4. Participant is positive for anti-citrullinated protein antibodies (ACPA).
5. Participant has a C-reactive protein (CRP) > upper limit normal (ULN) (5.0 g/L).
6. Participant has a negative tuberculosis test at Screening, defined as either negative QuantiFERON® test or purified protein derivative <5 mm of induration at 48 to 72 hours after the test was placed.

Exclusion Criteria:

1. Participant has Class IV RA according to ACR revised response criteria.
2. Participant has 1 or more significant concurrent medical conditions per investigator judgment, including but not limited to the following:

   * Poorly controlled diabetes or hypertension,
   * Chronic kidney disease stage IIIb, IV, or V,
   * Symptomatic heart failure according to New York Heart Association Classes II, III, or IV,
   * Myocardial infarction, unstable angina pectoris, stroke, or transient ischemic attack, within the past 12 months before randomization,
   * Severe chronic pulmonary disease, for example, requiring oxygen therapy,
   * Clinically significant hepatic diseases (i.e., hemochromatosis, Wilson's disease, alcoholic hepatitis, autoimmune liver disease, nonalcoholic steatohepatitis, or α-1-antitrypsin deficiency,
3. Participant has known history of prosthetic or native joint infection or human immunodeficiency virus or neurologic symptoms suggestive of central nervous system demyelinating disease.
4. Participant has a chronic inflammatory disease or connective tissue disease other than RA, including but not limited to; systemic lupus erythematosus, psoriatic arthritis, axial spondyloarthritis including ankylosing spondylitis and non radiographic axial spondylarthritis, reactive arthritis, gout, scleroderma, polymyositis, dermatomyositis and/or active fibromyalgia and/or multiple sclerosis.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-03 (Estimated); Primary Completion 2025-05 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants achieving clinical response according to the ACR 20 criteria at Week 12 | Baseline and Week 12
  Participants who met following 2 conditions for improvement from baseline were classified as meeting the ACR(American College of Rheumatology) 20 response criteria:
  * ≥ 20% improvement in 66-swollen joint count
  * ≥ 20% improvement in 68-tender joint count

SECONDARY OUTCOMES:
Clinical response at Week 12, assessed as the attainment of an LDA (Low Disease Activity) state defined | Baseline and Week 12
  * ACR 50 and ACR 70
  * DAS28-CRP < 3.2
  * CDAI (Clinical Disease Activity Index) ≤ 10
Clinical response at Week 12, assessed as remission defined | Baseline and Week 12
  * DAS28-CRP ≤ 2.6
  * CDAI ≤ 2.8
Improvement of physical function at Week 12 | Baseline and Week 12
  * ≥ 0.22 decrease in patient-reported ACR Core Set Values in participant's assessment of physical function using the HAQ-DI (Health Assessment Questionnaire - Disability Index)
  * <0.5 in participant's assessment of physical function using the HAQ-DI
Pain relief at Week 12 assessed by the (mean) change from Baseline | Baseline and Week 12
  - NRS-11 (11-point numeric scale)
Health-related quality of life at Week 12, assessed as the change from Baseline | Baseline and Week 12
  EuroQoL (EQ-5D-5L)

CONTACTS AND LOCATIONS:
Overall Officials: Jacob M. van Laar, MD, Principal Investigator — Department of Rheumatology & Clinical Immunology, University Medical Center Utrecht
Locations (1):
- University Medical Center Urtrecht, Utrecht, GA, Netherlands

IPD SHARING:
Plan to Share IPD: No